CLINICAL TRIAL: NCT01779453
Title: A Placebo-Controlled, Randomized, Double-Blind, Parallel Group, Drug Interaction Study to Evaluate the Safety, Tolerability and Effect on Atorvastatin Pharmacokinetics of ETC-1002 Added to Atorvastatin 10 mg/Day in Subjects With Hypercholesterolemia
Brief Title: A Study of the Safety, Pharmacokinetic Drug Interaction and Efficacy of ETC-1002 and Atorvastatin in Subjects With Hypercholesterolemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Esperion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1002-007
Record Dates: First submitted 2012-12-14; First posted 2013-01-30 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Hypercholesterolemia
Keywords: Atorvastatin; Drug-drug interaction; Combination therapy
MeSH Terms: conditions — Hypercholesterolemia | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ETC-1002 (Experimental): ETC-1002 treatment group, oral once daily
  Interventions: Drug: ETC-1002; Drug: Atorvastatin
- Placebo (Placebo Comparator): Placebo treatment group, oral once daily
  Interventions: Drug: Placebo; Drug: Atorvastatin

INTERVENTIONS:
Drug: ETC-1002 — Week 1-2, 60 mg/day; Week 3-4, 120 mg/day; Week 5-6, 180 mg/day; Week 7-8, 240 mg/day
  Arms: ETC-1002
Drug: Placebo — Placebo once daily for 8 weeks
  Arms: Placebo
Drug: Atorvastatin — Atorvastatin 10mg once daily for 8 weeks

SUMMARY:
This study will assess the safety, atorvastatin pharmacokinetics, and LDL-C lowering efficacy of ETC-1002 versus placebo in hypercholesterolemic subjects on background therapy of atorvastatin 10 mg.

ELIGIBILITY:
Inclusion Criteria:

* For subjects on current daily statin therapy - LDL-C 100-220 mg/dL and triglycerides <350 mg/dL (prior to switching to sponsor -provided atorvastatin 10 mg/day and stopping all other lipid-regulating drugs and supplements) at the S1 Visit,
* For subjects not on current daily statin therapy - LDL-C ≥ 110 mg/dL and ≤ 220 mg/dL

Exclusion Criteria:

* Acute significant cardiovascular disease
* Uncontrolled hypertension

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of atorvastatin and its active metabolites | 4 and 8 weeks
Peak plasma concentration (Cmax) of atorvastatin and its active metabolites | 4 and 8 weeks
Number of subjects with adverse events, clinical lab abnormalities and other safety findings | 8 weeks

SECONDARY OUTCOMES:
Percent change in LDL-C | 2, 4, 6 and 8 weeks
Percent change in other lipids and cardio-metabolic risk factors | 2, 4, 6 and 8 weeks

OTHER OUTCOMES:
Area under the plasma concentration versus time curve (AUC) and peak plasma concentration (Cmax) of ETC-1002 and its active metabolite | 4 and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Noah Rosenberg, MD, Study Director — Esperion Therapeutics, Inc.
Locations (3):
- United States (3):
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Richmond, Virginia